CLINICAL TRIAL: NCT06944626
Title: The Effect of Transcranial Direct Current Stimulation (tDCS) on Dyspnoea Perception, Pulmonary Function and Functional Level During COPD Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Istinye University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Assoc. Prof Dr, Okan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11/2024.K-73
Record Dates: First submitted 2025-03-23; First posted 2025-04-25 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: COPD; Dyspnea; tDCS
Keywords: COPD; tDCS; fNIRS; Dyspnea; Pulmonary function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Gruop (Experimental): Conventional physiotherapy + tDCS
  Interventions: Device: tDCS; Other: Conventional physiotherapy
- Sham group (Sham Comparator): Conventional physiotherapy + sham tDCS
  Interventions: Device: Sham tDCS; Other: Conventional physiotherapy

INTERVENTIONS:
Device: tDCS — tDCS will be applied to the dorsalateral prefrontal cortex with a current of 2 mA for 30 minutes on 3 consecutive days.
  Arms: Study Gruop
Device: Sham tDCS — The tDCS application will be increased to 2 mA for the first 30 seconds and will be reduced to 0 mA within 30 seconds after receiving current for 15 seconds. The electrodes will remain on the patient's head for the rest of the time (30 min in total).
  Arms: Sham group
Other: Conventional physiotherapy — Within the scope of conventional physiotherapy, respiratory control training, diaphragmatic breathing exercise, puckered lip breathing, relaxation exercises will be started 10 minutes after the start of tDCS or sham tDCS application.
  While tDCS or sham tDCS application continues, 10 repetitions will be performed in order and with time for rest between exercises.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a treatable disease characterized by irreversible and progressive airflow limitation, which is a cause of high morbidity and mortality. Dyspnea is an important component of COPD exacerbations that changes functional level and prognosis and limits the patient's quality of life and activities of daily living. Since COPD patients complain a lot of dyspnea associated with reduced exercise capacity and worsening lung function, there is a great need to develop effective physiologically based rehabilitation techniques to restore the dysfunctional respiratory motor system. Evidence supporting the importance of task-specific training based on neural plasticity also applies to pulmonary rehabilitation for COPD. Alterations in neuroplasticity and cortical excitability, tDCS is a promising technique for modulating brain activity. As a painless, easy-to-use and noninvasive technique, tDCS has shown efficacy in relieving pain, which shares the same neural substrates as dyspnea. Similarities have been established between the pathophysiology of dyspnea and pain. Close or even overlapping activation zones of brain structures involved in the integration of pain and dyspnea have been emphasized. Therefore, it is hypothesized that tDCS stimulation of areas where one or more of these cerebral structures are activated in pain may also have an effect on dyspnea. In light of this information, researchers believe that relieving dyspnea with tDCS will have an impact on the prognosis of patients during COPD exacerbations. In this context, researchers will evaluate the effects of tDCS on dyspnea perception, lung function, and functional level in patients with COPD exacerbation. When the literature was reviewed, no study on the use of tDCS in COPD patients was found. The use of tDCS as a non-invasive and easy-to-use effective treatment method with neuro-modulation to combat dyspnea and functional level in COPD patients constitutes the originality of the study.

Forty patients who were hospitalized in the Chest Diseases Service due to COPD exacerbation and met the inclusion criteria will be included in the study. The evaluation parameters included symptom assessment, breathlessness perception questionnaire, COPD assessment test, peripheral muscle strength assessment, grip strength assessment, pulmonary function test, Montreal cognitive assessment test, London chest activities of daily living scale, timed up and go test, hospital anxiety and depression scale, respiratory muscle strength, fNIRS and capnography. Assessments will take place before and after treatment. Sham (n:20) group will receive conventional physiotherapy and sham tDCS, while the Study (n:20) group will receive tDCS and conventional physiotherapy. For anodal tDCS, the anode electrode will be placed over the left primary motor cortex and the cathode will be placed over the right supraorbital region. For the study group, tDCS application will be applied with a current of 2 mA for 30 minutes on 3 consecutive days. In the sham group, tDCS application will be increased to 2 mA for the first 30 seconds and then decreased to 0 mA within 30 seconds after receiving current for 15 seconds. The electrodes will remain on the patient's head for the rest of the time (30 minutes in total).

In conclusion, the effects of tDCS on dyspnea perception, pulmonary function and functional level in COPD exacerbation period patients will be investigated. At the same time, the advantages of tDCS administration in COPD patients will be evaluated by examining its effects on cerebrovascular responses, tissue oxygenation, muscle strength, cognitive level, activity of daily living, anxiety and depression. It will provide different perspectives to clinicians and researchers who will create evaluation, treatment and study plans for COPD exacerbation period patients with limited treatment options and will be a guide for new research.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD and followed up for at least 6 months
* Hospitalised due to an exacerbation
* Have not taken any medication affecting the nervous system in the last 6 months
* Co-operative
* Have the ability to participate in working procedures
* Over 18 years of age,
* The specialist physician finds it suitable for physiotherapy applications,
* Volunteers who want to participate in the study

Exclusion Criteria:

* Having comorbidities other than COPD, such as bronchiectasis, lung cancer or asthma
* Surgery in the last 6 months (volume reduction surgery, etc.)
* Neuromuscular disease
* Pulmonary embolism or pulmonary oedema
* Presence of cranial, cardiac, spinal cord, intra-aural metal implants
* Epilepsy
* Patients on invasive mechanical ventilation
* Patient with cardiac pace maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Breathlessness Perception Questionnaire (BBQ): | Day 1 (before treatment) and day 3 (after treatment)
  The questionnaire consists of 11 items. Somatic focussing (BBQ-SF, 5 items) and activity avoidance (BBQ-AA, 6 items). Participants select a response for each item on a five-point scale from 'strongly disagree' (1 point) to 'strongly agree' (5 points), giving a total score between 11 and 55. A score of 11 reflects the absence of dyspnoea perception or dyspnoea-related kinesiophobia. High scores on the BBQ-SF reflect a perception that their illness is more harmful. High scores on the BBQ-AA reflect the patient's belief that physical activity that causes dyspnoea should be avoided as it may worsen their illness.
Oxygen saturation | Day 1 (before treatment) and day 3 (after treatment)
  The patient's oxygen saturation is measured by pulse oximetry.
COPD Assessment Test (CAT) | Day 1 (before treatment) and day 3 (after treatment)
  It is a one-dimensional scale consisting of 8 items that evaluates symptoms in COPD. It analyses the effect of symptoms such as cough, sputum, chest tightness, shortness of breath when climbing stairs, activity limitation at home, confidence when leaving home, sleep and energy on activities of daily living. Each question is numbered from 0 to 5 and the total score ranges from 0-40 points. The total score is classified according to five sections categorised according to the impact of symptoms on activities of daily living. According to this classification, the total score is categorised as follows: >30 points is considered as very high impact level, >20 points is considered as high impact level, 10-20 points is considered as medium impact level, <10 points is considered as low impact level, 5 points is considered as upper limit of normal impact level in healthy never smokers. The cut-off point for CAT in COPD was set as 10 points. Individuals will be asked to tick the most appropriate
Respiratory Muscle Strength | Day 1 (before treatment) and day 3 (after treatment)
  Respiratory muscle strength will be measured in accordance with the American Thoracic Society/European Respiratory Society (ATS/ERS) criteria using an intraoral pressure measuring device (MicroRPM, Micro Medical; UK). All measurements will be performed in sitting position. The nasal airway will be closed with a nose clip and a suitable mouthpiece will be used. For maximum inspiratory pressure (MIP), a maximal expiratory manoeuvre will be performed before the device is taken into the mouthpiece, followed by maximal inspiration (Müller manoeuvre) at maximum rate for 1-3 seconds. For maximum expiratory pressure (MEP), a maximum inspiratory manoeuvre will be performed before the device is taken into the mouth. This will be followed by maximal expiration (Valsalva manoeuvre) at maximum speed for 1-3 seconds. Three measurements will be repeated and the highest value will be recorded as cmH2O (ATS/ERS).
Functional Level Assessment | Day 1 (before treatment) and day 3 (after treatment)
  To assess the functional level of the patients, a 1 minute sit and stand test will be performed. The test, which is performed on a standard height (46) cm chair, will first be demonstrated by the physiotherapist. With the start command, the patients will be asked to switch from standing position to sitting without delay and repeat the test for 1 minute at the speed they determine and feel safe, in the form of full sitting and full standing. Care will be taken to ensure that the knee joint is in 90 degrees flexion when sitting and in full extension when standing.The number of times the person sits down and stands up during a minute will be recorded.
Near Infrared Spectroscopy (fNIRS): | Day 1 (before treatment) and day 3 (after treatment)
  fNIRS is a technique in which the amount of absorption of NIR light by chromophore molecules (such as oxy-Hb and deoxy-Hb, cytochrome-c oxidase (CCO), myoglobin) is measured as it passes through tissues. The changes in oxy- and deoxy-Hb are visualised with the inserted sensors. Two or more colours of light are used to differentially distinguish absorption changes due to oxy-/deoxy-Hb. These changes in blood concentration will be monitored online.Optodes will be placed in the bilateral prefrontal cortex.
Capnography | Day 1 (before treatment) and day 3 (after treatment)
  The capnograph is a monitoring device that provides a graphical continuous record (mmHg) of the CO2 concentration in expired gases during respiration, giving information about the number of breaths per minute and the amount of CO2 removed in each breath. It measures the partial pressure of CO2 in expired air, called ETCO2, a reliable and time-sensitive clinical measure of respiratory function. ETCO2 has good concurrent validity compared with direct blood measurements. This value of 35 mmHg and below is often used as a cut-off point to define hypocapnia.Measurement is performed with the help of a nasal cannula.
Dyspnoea assessment | Day 1 (before treatment) and day 3 (after treatment)
  Dyspnoea will be evaluated with Borg scale. The participant will be asked to tick a number between 0 and 10 on the scale for the severity of dyspnoea. 0 indicates no dyspnoea. 10 indicates very severe dyspnoea.
Heart rate | Day 1 (before treatment) and day 3 (after treatment)
  The patient's heart rate is measured by pulse oximetry.
Respiratory frequency | Day 1 (before treatment) and day 3 (after treatment)
  Respiratory frequency will be measured with a capnograph device.The capnograph is a monitoring device that provides a graphical continuous record (mmHg) of the CO2 concentration in expired gases during respiration, giving information about the number of breaths per minute and the amount of CO2 removed in each breath.
Modifiye Medical Research Council(MMRC) | Day 1 (before treatment) and day 3 (after treatment)
  It is an objective scale that evaluates dyspnoea, one of the most basic symptoms of COPD. It is a scale consisting of 5 items based on different levels of activities that may cause dyspnoea in daily life. There are activities with difficulty levels that may increase dyspnoea over 0-4 points. Individuals will tick the most appropriate statement among these statements.
Peak flow rate (PEF) | Day 1 (before treatment) and day 3 (after treatment)
  Measurement will be made with a spirometer. The test will start with inspiration-expiration at tidal volume. Then a deep inspiratory manoeuvre will be followed by a rapid expiration. Peak flow rate (PEF) will be recorded. The measured values will be expressed as a percentage of the expected values according to height, age, gender and body weight (Miller et al., 2005). PEF will be performed with a spirometer (Cosmed Pony FX, Italy) according to ATS/ ERS criteria. Appropriate sterilisation method recommended by the guideline, disposable, personalised mouthpieces and filters will be used against the risk of infection.
Forced expiratory volume in the first second (FEV1) | Day 1 (before treatment) and day 3 (after treatment)
  Measurement will be made with a spirometer. The test will start with inspiration-expiration at tidal volume. Then a deep inspiratory manoeuvre will be followed by a rapid expiration. Forced expiratory volume in the first second (FEV1) will be recorded. The measured values will be expressed as a percentage of the expected values according to height, age, gender and body weight (Miller et al., 2005). FEV1 will be performed with a spirometer (Cosmed Pony FX, Italy) according to ATS/ ERS criteria. Appropriate sterilisation method recommended by the guideline, disposable, personalised mouthpieces and filters will be used against the risk of infection.
Forced vital capacity (FVC) | Day 1 (before treatment) and day 3 (after treatment)
  Measurement will be made with a spirometer. The test will start with inspiration-expiration at tidal volume. Then a deep inspiratory manoeuvre will be followed by a rapid expiration. Forced vital capacity (FVC) will be recorded. The measured values will be expressed as a percentage of the expected values according to height, age, gender and body weight (Miller et al., 2005). FVC will be performed with a spirometer (Cosmed Pony FX, Italy) according to ATS/ ERS criteria. Appropriate sterilisation method recommended by the guideline, disposable, personalised mouthpieces and filters will be used against the risk of infection.
FEV1/FVC | Day 1 (before treatment) and day 3 (after treatment)
  Measurement will be made with a spirometer. The test will start with inspiration-expiration at tidal volume. Then a deep inspiratory manoeuvre will be followed by a rapid expiration. FEV1/FVC will be recorded. The measured values will be expressed as a percentage of the expected values according to height, age, gender and body weight (Miller et al., 2005). FEV1/FVC will be performed with a spirometer (Cosmed Pony FX, Italy) according to ATS/ ERS criteria. Appropriate sterilisation method recommended by the guideline, disposable, personalised mouthpieces and filters will be used against the risk of infection.
Fatigue assessment | Day 1 (before treatment) and day 3 (after treatment)
  Fatigue will be assessed using the Borg scale. The participant will be asked to mark a number between 0 and 10 on the Borg scale for the severity of fatigue. 0 indicates no fatigue. 10 indicates very severe fatigue.

SECONDARY OUTCOMES:
Peripheral Muscle Strength Assessment | Day 1 (before treatment) and day 3 (after treatment)
  Peripheral muscle strength of the shoulder abductor and flexor, elbow flexor, wrist extensor, knee extensor, hip flexor and ankle dorsiflexor muscles will be measured with a portable manual muscle strength measuring device (Model 01165, Lafayette, IN, USA). Measurements will be repeated three times for the right and left side.
Montreal Cognitive Assessment Test (MoCA) | Day 1 (before treatment) and day 3 (after treatment)
  It is a questionnaire developed to evaluate cognitive functions. The cognitive functions assessed are concentration, language, memory, orientation, abstract thinking, visual structuring, calculation and executive functions. The maximum score that can be obtained from the test is 30, 21 or above indicates the absence of mild cognitive impairment.
London Chest Activities of Daily Living Scale (LCADL) | Day 1 (before treatment) and day 3 (after treatment)
  It will be used for the assessment of activities of daily living. With 15 questions, the questionnaire questions the severity of dyspnoea during activities of daily living and includes sub-items such as domestic activities, leisure time, self-care and physical activities. Each item will be scored between 0 and 5. A high score indicates inadequacy in activities of daily living. The maximum total score is 75.

CONTACTS AND LOCATIONS:
Locations (1):
- İstinye Üniversitesi, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided